CLINICAL TRIAL: NCT05664217
Title: A Phase 2/3, Randomized, Double Blind, Placebo-controlled, Multicenter Study of NKTR-255 vs Placebo Following CD19-directed CAR-T Cell Therapy in Patients With Relapsed/Refractory Large B-cell Lymphoma
Brief Title: NKTR-255 vs Placebo Following CD19-directed CAR-T Therapy in Patients With Relapsed/Refractory Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to end the study
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-255-01
Record Dates: First submitted 2022-12-01; First posted 2022-12-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Non-Hodgkin Lymphoma; Relapsed/Refractory Diffuse Large B-cell Lymphoma
Keywords: NHL; LBCL; DLBCL; CAR; CAR-T; cell therapy; NKTR-255; chimeric antigen receptor; autologous T-cell; axi-cel; liso-cel; immunotherapy; B-cell malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: The study is conducted in two stages, with routine safety monitoring being conducted by the Data Monitoring Committee (DMC) on a regular basis. An enrollment pause will be implemented at the end of Stage 1, and the DMC will review safety and efficacy data from all available cohorts to make go/no-go and dose selection recommendations for Stage 2. The study team will be unblinded at the end of Stage 1 to review totality of the data including efficacy, safety, PK, and PD data.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study. The Investigator, the patients, and all study site and Nektar personnel involved in study activities, other than those involved in dispensing the study drugs, conducting PK, PD sample analyses, and personnel supporting unblinded monitoring for drug accountability, must remain blinded to each patient's treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stage 1 NKTR-255 at 1.5 µg/kg (Experimental): In this arm of Stage 1 (Phase 2 of the study), NKTR-255 will be dosed at 1.5 µg/kg. NKTR-255 will be administered intravenously approximately 14 days after CD19-directed CAR-T cell infusion.
  Patients will be dosed every 3 weeks for up to 7 cycles or 5 months, whichever is earlier, in the absence of disease progression or unacceptable toxicity.
  The dose regimen for Stage 2 (Phase 3 of the study) will be selected based on the results of Stage 1 as reviewed by the Data Monitoring Committee (DMC) and the study team.
  Interventions: Drug: NKTR-255 at 1.5 µg/kg
- Stage 1 NKTR-255 at 3.0 μg/kg (Experimental): In this arm of Stage 1 (Phase 2 of the study), NKTR-255 will be dosed at 3.0 μg/kg. NKTR-255 will be administered intravenously approximately 14 days after CD19-directed CAR-T cell infusion.
  Patients will be dosed every 3 weeks for up to 7 cycles or 5 months, whichever is earlier, in the absence of disease progression or unacceptable toxicity.
  The dose regimen for Stage 2 (Phase 3 of the study) will be selected based on the results of Stage 1 as reviewed by the Data Monitoring Committee (DMC) and the study team.
  Interventions: Drug: NKTR-255 at 3.0 μg/kg
- Stage 1 NKTR-255 at 3.0/6.0 μg/kg (Experimental): In this arm of Stage 1 (Phase 2 of the study), patients will be dosed with 3.0 μg/kg NKTR-255 in Cycle 1 (C1) and continue in Cycle 2 and subsequent cycles (C+) with 6.0 μg/kg NKTR-255 (hereinafter referred to as 3.0/6.0 µg/kg NKTR-255).
  NKTR-255 will be administered intravenously approximately 14 days after CD19-directed CAR-T cell infusion.
  Patients will be dosed every 3 weeks for up to 7 cycles or 5 months, whichever is earlier, in the absence of disease progression or unacceptable toxicity.
  The dose regimen for Stage 2 (Phase 3 of the study) will be selected based on the results of Stage 1 as reviewed by the Data Monitoring Committee (DMC) and the study team.
  Interventions: Drug: NKTR-255 at 3.0/6.0 μg/kg
- Placebo (Placebo Comparator): Placebo is commercially available 0.9% Sodium Chloride Solution for Injection (USP). Placebo will be administered intravenously approximately 14 days after CD19-directed CAR-T cell infusion. Placebo will be infused every 3 weeks for up to 7 cycles or 5 months, whichever is earlier.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: NKTR-255 at 1.5 µg/kg — NKTR-255 at 1.5 µg/kg
  Other Names: Polymer-conjugated interleukin (IL)-15 Receptor Agonist
  Arms: Stage 1 NKTR-255 at 1.5 µg/kg
Drug: NKTR-255 at 3.0 μg/kg — NKTR-255 at 3.0 μg/kg
  Other Names: Polymer-conjugated interleukin (IL)-15 Receptor Agonist
  Arms: Stage 1 NKTR-255 at 3.0 μg/kg
Drug: NKTR-255 at 3.0/6.0 μg/kg — NKTR-255 at 3.0/6.0 μg/kg
  Other Names: Polymer-conjugated interleukin (IL)-15 Receptor Agonist
  Arms: Stage 1 NKTR-255 at 3.0/6.0 μg/kg
Other: Placebo Comparator — Commercially available 0.9% Sodium Chloride Solution for Injection (USP)
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of NKTR-255 following CD19-directed chimeric antigen (CAR)-T cell therapy in patients with relapsed or refractory (R/R) large B-cell lymphoma (LBCL).

NKTR-255 is an investigational IL-15 receptor agonist designed to boost the immune system's natural ability to fight cancer. T cells are infection fighting blood cells that can kill tumor cells. Chimeric antigen (CAR)-T cell product consists of genetically engineered T-cells, modified to recognize CD19, a protein on the surface of cancer cells. These CD19-specific T cells may help the body's immune system identify and kill CD19-positive cancer cells. Giving NKTR-255 following the treatment with CD19 CAR-T cell therapy may work better in treating large B-cell lymphoma than either drug alone.

DETAILED DESCRIPTION:
Patients will be treated with lymphodepletion chemotherapy (as recommended by the CAR-T cell manufacturer) and soon after will receive a one-time CD19-directed CAR-T cell infusion (as per product label). Study drug (NKTR-255 or placebo) will be administered intravenously approximately 14 days after CAR-T cell infusion and administered every 3 weeks for up to 7 cycles or 5 months (whichever is earlier) in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients will be followed-up at 30 days, and then at 9,12,18, 24, and 36 months after CAR-T cell infusion.

The Stage 1 (Phase II) portion of the study only enrolled to the dose optimization. Primary endpoint data will be available in the second half of 2024.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female ≥ 18 years of age at the time of consent.
2. Received standard of care therapy with axi-cel or liso-cel (Stage 1 and Stage 2), or tisa-cel (Stage 2 only), for the respective FDA (or Summary of Product Characteristics [SmPC]) approved indication(s):

   1. liso-cel: Patients with LBCL (including diffuse LBCL [DLBCL] not otherwise specified [including DLBCL arising from indolent lymphoma], high-grade B-cell lymphoma, primary mediastinal LBCL, and follicular lymphoma Grade 3B), who have:

      1. refractory disease to first-line chemoimmunotherapy or relapse within 12 months of first-line chemoimmunotherapy;
      2. refractory disease to first-line chemoimmunotherapy or relapse after first-line chemoimmunotherapy and are not eligible for hematopoietic stem cell transplantation (HSCT) due to comorbidities or age; or,
      3. relapsed or refractory disease after two or more lines of systemic therapy.
   2. axi-cel: For the treatment of adult patients with LBCL that is:

      1. refractory to first-line chemoimmunotherapy;
      2. relapses within 12 months of first-line chemoimmunotherapy; or
      3. R/R LBCL after 2 lines of systemic therapy, including DLBCL not otherwise specified, primary mediastinal LBLC, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma.
   3. tisa-cel (Stage 2 only): Adult patients with R/R LBLC after two lines of systemic therapy including DLBCL not otherwise specified, high grade B-cell lymphoma and DLBCL arising from follicular lymphoma.
3. Received lymphodepleting chemotherapy regimen according to the respective FDA (or SmPC) label for CAR-T cell therapy.
4. Fluorodeoxyglucose (FDG)-avid disease on positron emission tomography (PET) imaging within 30 days prior to CAR-T cell infusion.
5. FDG avid lesion(s) on PET/computed tomography (CT) scan following bridging therapy and prior to lymphodepletion, where applicable.
6. Evidence of CD19 expression on any prior or current NHL tumor specimen or a high likelihood of CD19 expression based on disease histology per investigator's assessment.
7. Within 7 days prior to leukapheresis, patient should have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1 (Appendix 3).
8. Regarding prior systemic anti-tumor therapy:

   1. At least 3 months have elapsed since systemic immune checkpoint inhibitory/immune stimulatory therapy (eg, ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc).
   2. At least 2 weeks have elapsed since other prior systemic antitumor therapy.
   3. Bridging therapy (including steroids) is permitted between leukapheresis and lymphodepletion as long as Exclusion Criterion 1 is satisfied.
9. Adequate organ function, defined as:

   1. Adequate bone marrow function (prior to lymphodepletion) for lymphodepletion chemotherapy defined as: absolute neutrophil count (ANC) ≥ 1000 cells/mm3, platelets ≥ 50,000 cells/mm3, and hemoglobin ≥ 8 g/dL in the absence of bone marrow involvement by lymphoma. No transfusion within 3 days of bone marrow function assessment; growth factor support is allowed as per institutional practice.
   2. Calculated creatinine clearance (Cockcroft/Gault) > 30 mL/min (Appendix 4).
   3. ALT and AST ≤ 3 × upper limit of normal (ULN; or < 5 × ULN for patients with lymphomatous infiltration of the liver) and total bilirubin ≤ 2 × ULN (or < 3.0 × ULN for patients with Gilbert's syndrome or lymphomatous infiltration of the liver).
   4. Adequate pulmonary function, oxygen saturation on room air (SaO2) ≥ 92%. Patients with a history of interstitial lung disease should undergo pulmonary function testing and must have a forced expiratory volume in 1 second (FEV1) of ≥ 50% of predicted value or diffusing capacity of the lung for carbon monoxide (DLCO; corrected) ≥ 40% of predicted value.
   5. Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) ≥ 40% as assessed by echocardiogram (ECHO) or multiple uptake gated acquisition (MUGA) within 60 days before randomization.
10. ECG demonstrating Fridericia's corrected QT interval (QTcF) < 470 ms. Patients with QTcF ≥ 470 ms will require clearance by a local cardiologist.
11. Women of reproductive potential (defined as all women physiologically capable of becoming pregnant) must agree to use suitable methods of contraception from the start of study treatment until 1 month after the last dose of study drug (Appendix 6).
12. Males who have partners of reproductive potential must agree to use an effective barrier contraceptive method from the start of study treatment until 1 month after the last dose of study drug.
13. Ability to understand and provide written informed consent.
14. Able and willing to comply with study visit schedule and procedures, including tumor biopsy where accessible.

    Additional Eligibility Criteria Following CD19 Targeted CAR-T Cell Infusion

    Patients who have received commercially released CAR-T cell infusion must satisfy the following criteria on the day of randomization:
15. No fever ≥ 38.0°C/Grade ≥ 1 CRS (American Society for Transplant and Cellular Therapy [ASTCT] criteria within 24 hours.
16. No Grade ≥ 3 CRS (ASTCT criteria) within 72 hours.
17. No previous Grade ≥ 3 immune effector cell-associated neurotoxicity syndrome (ICANS) of > 72 hours duration.
18. No Grade ≥ 2 ICANS (ASTCT criteria).
19. No tocilizumab and/or dexamethasone within 48 hours.
20. No active, serious, and/or uncontrolled infection(s).
21. No other contraindication according to the Investigator's assessment.
22. Patients must satisfy the following laboratory test results:

    * ANC or absolute granulocyte count (AGC) ≥ 1000/μL
    * Platelets ≥ 30,000/μL
    * Hemoglobin ≥ 8 g/dL
    * Leukocytes ≥ 3000/μL Randomization should occur no more than 1 day before the first study drug infusion.

Exclusion Criteria:

1. Use of therapeutic doses of corticosteroids (≥ 5 mg/day prednisone or equivalent) or other systemic immunosuppression within 7 days prior to leukapheresis or within 72 hours prior to CAR-T cell infusion. Topical and/or inhaled steroids are permitted.
2. Prior treatment with any CD19-directed CAR-T cell therapy other than the treatment planned per Inclusion Criterion 2.
3. For allogeneic hematopoietic cell transplant recipients, active graft versus host disease (GVHD) and/or systemic GVHD therapy during screening or up to 30 days prior to leukapheresis.
4. Known active hepatitis B (detectable hepatitis B DNA) or hepatitis C (detectable hepatitis C RNA).
5. Known human immunodeficiency virus (HIV) infection.
6. Pregnant or breastfeeding women.
7. Prior treatment with any IL-2 or IL-15 agonist and/or biosimilar agents.
8. Active autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, ulcerative colitis, Crohn's disease], celiac disease, or other serious chronic gastrointestinal conditions associated with diarrhea, autoimmune vasculitis, systemic lupus erythematosus, Wegener syndrome [granulomatosis with polyangiitis], myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.) within 1 year prior to randomization. The following are exceptions to this criterion:

   1. Vitiligo
   2. Alopecia
   3. Hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
   4. Type 1 diabetes mellitus
   5. Psoriasis not requiring systemic treatment
   6. Conditions considered to be low risk of serious deterioration by the Investigator and with Medical Monitor approval
9. History of any one of the following cardiovascular conditions within the 6 months prior to randomization: class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, or unstable angina; unless clearance by a cardiologist is obtained. History of other clinically significant cardiac disease that, in the opinion of the Investigator or designee, is a contraindication to study treatment is also excluded.
10. History or presence of clinically relevant central nervous system (CNS) pathology, such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, or psychosis that in the opinion of the Investigator is a contraindication to study treatment.
11. History of CNS lymphoma, primary CNS lymphoma, brain metastases, or detectable malignant cells in the cerebrospinal fluid.
12. History of solid organ transplantation.
13. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the Medical Monitor.
14. Presence of any indwelling line or drain (eg, percutaneous nephrostomy tube, indwelling foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted.
15. Active or current participation on any other interventional studies.
16. Use of an investigational agent or an investigational device within 28 days of CAR-T cell therapy.
17. Live, attenuated vaccines are prohibited within 30 days of randomization.
18. Any condition including medical, emotional, psychiatric, or logistical that, in the opinion of the Investigator, would preclude the patient from adhering to the protocol or would increase the risk associated with study participation or study drug administration or interfere with the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate at month 6 | At month 6 after the first infusion with study drug
  The incidence of complete response by the Lugano Classification (Cheson et al, 2014) as determined by blinded independent central review (BICR)
Event-free survival (EFS) | Up to 3 years after the first infusion with study drug
  Event-free survival is defined as the time from randomization to the earliest date of disease progression by the Lugano Classification (Cheson et al, 2014) as determined by BICR, commencement of new lymphoma therapy, or death from any cause.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) and laboratory abnormalities by type and severity. | From the first dose of study drug up to 30 days after the last dose of study drug
  Incidence of treatment-emergent adverse events and significant laboratory abnormalities using Medical Dictionary for Regulatory Activities (MedDRA) for characterizing reported events and central laboratory references ranges for abnormal laboratory values. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria (Lee 2019). Other AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 (CTCAE 2017).
Complete response (CR) rate at month 3 | At month 3 after the first infusion with study drug
  The incidence of complete response at month 3 by the Lugano Classification (Cheson et al, 2014) as determined by blinded independent central review (BICR)
Best overall Complete response (CR) rate | Up to 3 years
  The incidence of complete response in study by the Lugano Classification (Cheson et al, 2014) as determined by blinded independent central review (BICR)
Objective response rate (ORR) at month 3 | At month 3 after the first infusion with study drug
  The incidence of objective response rate is defined as the incidence of either a complete response or a partial response by the Lugano Classification (Cheson et al, 2014) as determined by BICR
Objective response rate (ORR) at month 6 | At month 6 after the first infusion with study drug
  The incidence of objective response rate is defined as the incidence of either a complete response or a partial response by the Lugano Classification (Cheson et al, 2014) as determined by BICR
Best overall objective response rate (ORR) | Up to 3 years
  The incidence of objective response rate in study is defined as the incidence of either a complete response or a partial response by the Lugano Classification (Cheson et al, 2014) as determined by BICR
Duration of Response (DOR) | Time Frame: Up to 3 years
  The duration of response is derived only among subjects who experience an objective response per Lugano Classification (Cheson et al, 2014) as determined by blinded central review and is defined as the time from first response to disease progression per the Lugano Classification or death from any cause
Progression-Free Survival (PFS) | Up to 3 years
  Progression Free Survival is defined as the time from randomization to disease progression per Lugano Classification (Cheson et al, 2014) or death from any cause
Overall Survival (OS) | Up to 3 years
  Overall survival is defined as the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (22):
- United States (22):
  - University of California San Diego, La Jolla, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University Of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Fairway, Kansas
  - University of Maryland, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute - Winston-Salem, Winston-Salem, North Carolina
  - Oncology Hematology Care Inc - Cincinnati, Cincinnati, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - Fred Hutchinson/University of Washington, Seattle, Washington